CLINICAL TRIAL: NCT06359379
Title: Phase 2 Study of Ropidoxuridine as a Radiation Sensitizing Agent During Radiotherapy in Patients With Newly Diagnosed IDH-Wildtype Glioblastoma With Unmethylated MGMT Promoter
Brief Title: Ropidoxuridine as a Radiosensitizer in Newly Diagnosed IDH-Wildtype Glioblastoma With Unmethylated MGMT Promoter
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to the sponsor's decision.
Sponsor: Shuttle Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S22-11168
Record Dates: First submitted 2024-03-24; First posted 2024-04-11 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Glioblastoma, IDH-wildtype
Keywords: radiotherapy; radiation sensitizing agent; ropidoxuridine; unmethylated MGMT promoter
MeSH Terms: conditions — Glioblastoma | interventions — ropidoxuridine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ropidoxuridine 960 mg (Experimental): Ropidoxuridine is administered orally at 960 mg, 5 days a week for a total of 7 weeks, starting 1 week before the initiation of radiotherapy.
  Interventions: Drug: Ropidoxuridine
- Ropidoxuridine 1200 mg (Experimental): Ropidoxuridine is administered orally at 1200 mg, 5 days a week for a total of 7 weeks, starting 1 week before the initiation of radiotherapy.
  Interventions: Drug: Ropidoxuridine

INTERVENTIONS:
Drug: Ropidoxuridine — Ropidoxuridine is administered daily, 5 days a week, for 7 weeks, starting one week prior to radiotherapy, and then concurrently with a standard 60 Gy radiotherapy, followed by a 4-week rest period.
  Other Names: 5-iodo-2-pyrimidinone-2'-deoxyribose

SUMMARY:
This is a randomized, open-label, phase 2 study evaluating the safety and efficacy of oral ropidoxuridine as a radiation-sensitizing agent in patients with newly diagnosed wild-type isocitrate dehydrogenase glioblastoma with an unmethylated O6-methylguanine-DNA methyltransferase promoter, undergoing standard 60 Gy radiotherapy.

DETAILED DESCRIPTION:
This is a randomized, open-label phase 2 study to assess the safety and efficacy of oral ropidoxuridine as a radiation sensitizing agent in patients with newly diagnosed wildtype isocitrate dehydrogenase glioblastoma with unmethylated O6-methylguanine-DNA methyltransferase promoter, receiving standard 60 Gy radiotherapy.

In the dose optimization phase, a group of 40 patients will be evenly divided, with a 1:1 randomization, to receive ropidoxuridine for a duration of 7 weeks. They will be administered daily ropidoxuridine at two dose levels: either 960 mg or 1200 mg. This administration will occur 5 days a week, from Monday to Friday. Treatment with ropidoxuridine will start one week before radiotherapy (induction period) and continue concomitantly with 60 Gy standard radiotherapy fractionated in 2 Gy daily doses (Monday through Friday weeks 2 to 7, treatment period)), followed by a 4-week rest period. Following completion of this 11-week active study period, maintenance therapy, including temozolomide, tumor treating field device (Optune®), or other available treatment modalities, may be initiated at the discretion of the Investigator.

Analysis of the pharmacokinetic, safety and tolerability data for the two cohorts will determine the optimal dose of ropidoxuridine, to be administered to the next cohort of 14 patients for determination of efficacy, compared to historical controls.

A magnetic resonance imaging ( MRI) will be performed at the end of the active study period (Week 11). This MRI should not be used for disease assessment due to increased contrast enhancement in the acute radiation reaction phase, unless there is evidence of progression outside the radiotherapy fields. Radiographic disease assessment will be performed in accordance with community standard of care guidelines, every 3 months until disease progression. After the confirmed disease progression, survival monitoring follow-ups will occur every three months.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent form signed and dated by patient or legally authorized representative according to local guidelines, prior to the performance of any study-specific procedures, sampling, or analyses. Participants with impaired decision-making capacity must have a close caregiver or legally authorized representative present.
* Histologically confirmed supratentorial glioblastoma isocitrate dehydrogenase (IDH) wild-type classification (2021 World Health Organization Classification of Tumours, 5th Edition, Volume 6) with unmethylated O6-methylguanine-DNA-methyltransferase (MGMT) promoter (defined as MGMT methylation status ≤20% by pyrosequencing, and no prior radiation, electric field, or systemic therapy. Glucocorticoid therapy for symptom control is allowed.
* Patients should, in the opinion of the investigator, be candidates for 60 Gy radiotherapy in 2 Gy fractions over 6 weeks, per standard of care. Hypofractionated radiotherapy schedules (e.g., 36 Gy in 3 Gy fractions) are not allowed.
* Eastern Cooperative Oncology Group performance status of 0, 1 or 2.
* Adequate renal, liver and bone marrow function:

  * Hemoglobin >9.0 g/dL
  * Absolute neutrophil count >1.5 × 10^9/L
  * Platelet count >100 × 10^9/L
  * Total bilirubin ≤1.5 × upper limit of normal (ULN), unless due to documented Gilbert's disease (≤3 × ULN)
  * Aspartate aminotransferase / alanine aminotransferase ≤4×ULN
  * Creatinine clearance ≥60 mL/min calculated as per Cockcroft-Gault equation.
* Life expectancy ≥12 weeks.
* Have recovered from the immediate post-operative period and is maintained on a stable corticosteroid regimen (no increase for 5 days) prior to initiation of study treatment.
* Female patients, of childbearing potential, must have a negative serum pregnancy test within 7 days prior to taking study medication and agree to use at least one highly effective form of contraception during study treatment and for at least 120 days after the last dose of study treatment.
* Male patients must agree to use an adequate method of contraception from enrollment through 120 days after the last dose of study treatment.

Exclusion Criteria:

* Any prior treatment for glioblastoma, including chemotherapy, immunotherapy, targeted therapy or therapy with biologic agent (including immunotoxins, immunoconjugates, antisense, peptide receptor antagonists, interferons, interleukins, lymphokine-activated killer cell therapy or gene therapy), or radiotherapy. Glucocorticoid therapy is permitted.
* Second primary malignancy expected to require active treatment within a 6-month period (except basal cell or early-stage squamous cell carcinoma of the skin that may be excised). Patients who had another malignancy in the past but have been free of active disease for more than 1 year, are eligible even if under active surveillance, at the discretion of the Investigator. Adjuvant anti hormonal treatment for prior breast or prostate cancer is allowed, but no other concomitant anticancer treatment.
* Any investigational therapy (for any concomitant condition) within 28 days or within 5 half-lives of study entry (whichever is shorter).
* Use of acid-reducing agents including proton pump inhibitors and histamine-2 blockers.
* Inability to comply with protocol or study procedures.
* Women who are pregnant or breastfeeding.
* Inability to swallow oral medication or gastrointestinal disorder expected to severely affect drug absorption (e.g., short bowel syndrome).
* Ongoing bacterial, viral, or fungal infection requiring systemic therapy. Prophylactic therapy is allowed. Patients with a history of Human Immunodeficiency Virus, Hepatitis B virus, Hepatitis C virus infection are allowed if treated with effective anti-viral therapy that results in undetectable viral load.
* Any medical condition, which in the opinion of the Investigator, places the patient at an unacceptably high risk for toxicities, or makes the patient unsuitable for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-09-02 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Number of patients treated with oral ropidoxuridine at dose levels of 960 and 1200 mg once daily, with treatment-related adverse events assessed by CTCAE v5.0. | From the first day of treatment start until 30 days after treatment completion
adiographic response rate, disease control rate, best overall response, and duration of overall response in patients treated with oral ropidoxuridine at 960 and 1200 mg daily doses, assessed using the Response Assessment in Neuro-Oncology criteria. | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months.
Maximum plasma concentration for orally administered ropidoxuridine, at dose levels of 960 and 1200 mg once daily. | he first 36 days of treatment.
Trough plasma concentration of orally administered ropidoxuridine, at dose levels of 960 and 1200 mg once daily | The first 36 days of treatment.
Time to maximum plasma concentration for orally administered ropidoxuridine, at dose levels of 960 and 1200 mg once daily. | The first 36 days of treatment.
Area under the curve for orally administered ropidoxuridine, at dose levels of 960 and 1200 mg once daily. | The first 36 days of treatment.
Half-life for orally administered ropidoxuridine, at dose levels of 960 and 1200 mg once daily. | The first 36 days of treatment.

SECONDARY OUTCOMES:
Overall survival at 12 months | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months.
Radiographic Response Rate | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months.
Disease Control Rate | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months.
Best Overall Response | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months.
Duration of Response | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months.
Overall Survival | From date of randomization until the date of death from any cause, whichever came first, assessed up to 100 months.
Progression-Free Survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months.
Six-Month Progression-Free Survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 6 months.
Fraction of patients with tumor progression outside of the treatment area. | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months.
Quantification of 9 relevant neurologic domains based on the NANO scale. | Measured from the time of study enrollment until 28 (±7) days following the completion of study treatment.
  The Neurologic Assessment in Neuro-Oncology (NANO) scale is a clinical tool used to measure neurological function in patients with brain tumors. The scale can range from a score of 0 to a maximum score that depends on the severity and number of deficits. Higher scores on the NANO scale typically indicate a greater degree of neurological impairment.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - Miami Cancer Institute, Miami, Florida
  - John Theurer Cancer Center at the Hackensack University Medical Center, Hackensack, New Jersey
  - Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Virginia, Charlottesville, Virginia